

# **Trial Statistical Analysis Plan**

c13209134 -01

**BI Trial No.:** 1237.34 Post-marketing surveillance (PMS) on long-term use of Title: tiotropium+olodaterol fixed dose combination (Tio+Olo FDC) 5μg/5μg in patients with chronic obstructive pulmonary disease (chronic bronchitis, emphysema) in Japan. Including Protocol Amendment c02840643-02. Investigational Tiotropium+olodaterol fixed dose combination solution for **Product(s):** inhalation -RESPIMAT Responsible trial statistician(s): Address: Phone: , Fax: **Date of statistical** 29 Nov 2018 SIGNED analysis plan: Version: Final **** 

Proprietary confidential information

© 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1237.34 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **TABLE OF CONTENTS** 1.

| TITLE | PAGE | 1 |
|--------|------------------------------------------------|----|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | OF TABLES | 3 |
| 2. | LIST OF ABBREVIATIONS | 4 |
| 3. | INTRODUCTION | 6 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | 7 |
| 5. | ENDPOINT(S) | 8 |
| 5.1 | PRIMARY ENDPOINT(S) | |
| 5.2 | SECONDARY ENDPOINT(S) | |
| 5.2.1 | Key secondary endpoint(s) | |
| 5.2.2 | Secondary endpoint(s) | |
| 5.3 | FURTHER ENDPOINT(S) | |
| 5.4 | OTHER VARIABLE(S) | |
| 6. | GENERAL ANALYSIS DEFINITIONS | 12 |
| 6.1 | TREATMENT(S) | |
| 6.2 | IMPORTANT PROTOCOL VIOLATIONS | |
| 6.3 | PATIENT SETS ANALYSED | |
| 6.5 | POOLING OF CENTRES | 13 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| 6.7 | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| 7. | PLANNED ANALYSIS | 15 |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | 15 |
| 7.3 | TREATMENT COMPLIANCE | 15 |
| 7.4 | PRIMARY ENDPOINT(S) | 15 |
| 7.5 | SECONDARY ENDPOINT(S) | |
| 7.5.1 | Key secondary endpoint(s) | 16 |
| 7.5.2 | (Other) Secondary endpoint(s) | 16 |
| 7.7 | EXTENT OF EXPOSURE | 16 |
| 7.8 | SAFETY ANALYSIS. | 16 |
| 7.8.1 | Adverse events | |
| 7.8.2 | Laboratory data | |
| 7.8.3 | Vital signs | |
| 7.8.4 | ECG | |
| 7.8.5 | Others | |
| 8. | REFERENCES | 19 |
| • | | |
| 10. | HISTORY TABLE | 21 |

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1237.34 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# List of Tables

| Table 6.2:1 Important protocol violations | .12 |
|----------------------------------------------------------|------|
| Table 6.7:1 Baseline, time windows and calculated visits | . 14 |
| Table 10:1 History table | .21 |

TSAP for BI Trial No: 1237.34 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

Include a list of all abbreviations used in the TSAP

| Definition / description |
|------------------------------------------------------------|
| Adverse Drug Reaction |
| Adverse event |
| Blinded report planning meeting |
| COPD Assessment Test |
| Chronic Obstructive Pulmonary Disease |
| Case Report Form |
| Clinical Trial Report |
| Boehringer Ingelheim Data Management and Statistics Manual |
| Drug Regulatory Affairs |
| Dictionary Maintenance Group |
| Forced Expiratory Volume in one second |
| Forced Vital Capacity |
| Inhaled Corticosteroid |
| Long Acting Beta2 Agonist |
| Long Acting Muscarinic Antagonist |
| Last observation carried forward |
| Medical Dictionary for Regulatory Activities |
| Medical Quality Review Meeting |
| Non-interventional Study |
| Patient's Global Rating |
| Project Statistician |
| Pulmonary Function Test |
| Preferred term |
| Protocol violation |
| Lower quartile |
| Upper quartile |
| Statistical analysis |
| Serious Adverse Event |

Boehringer Ingelheim
TSAP for BI Trial No: 1237.34
Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|------|---------------------------------------|
| SADR | Serious Adverse Drug Reaction |
| SD | Standard deviation |
| SMQ | Standardised MedDRA query |
| SOC | System organ class |
| TCM | Trial Clinical Monitor |
| TESS | Treatment emergent signs and symptoms |
| ToC | Table of contents |
| TMW | Trial Medical Writer |
| TSAP | Trial statistical analysis plan |

## 3. INTRODUCTION

The purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the post-marketing surveillance (PMS) data.

This TSAP assumes familiarity with the Non-interventional Study Protocol (NIS Protocol), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in NIS Protocol Section 9.7 "DATA ANALYSIS". Therefore, TSAP readers may consult the NIS Protocol for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size.

SAS® Version 9.4 or later will be used for all analyses.

TSAP for BI Trial No: 1237.34 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

No change has been made in the planned analyses from the statistical methods described in the NIS Protocol.

TSAP for BI Trial No: 1237.34

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 5. ENDPOINT(S)

#### 5.1 PRIMARY ENDPOINT(S)

There is no primary endpoint for effectiveness the primary objective of the PMS study is the evaluation of safety (see the NIS Protocol Section 9.1).

## 5.2 SECONDARY ENDPOINT(S)

#### 5.2.1 Key secondary endpoint(s)

This section is not applicable as no key secondary endpoint has been specified in the protocol.

#### 5.2.2 Secondary endpoint(s)

The secondary endpoints will be used as defined in the NIS Protocol Section 9.1

## 5.3 FURTHER ENDPOINT(S)

The other endpoints will be used as stated in the NIS Protocol Section 9.1.

## 5.4 OTHER VARIABLE(S)

Demographic data and baseline characteristics:

- Gender: male, female
- Age [years]
  - Age [years] = Actual age based on the first administration of Spiolto Respimat
- Age class1 [years]: <65, >=65
- Age class2 [years]: <65, 65 to <75, >=75
- Height [cm]
- Weight [kg]
- Weight class [kg]: <50, 50 to <70, >=70
- Body mass index (BMI) [kg/m<sup>2</sup>] BMI [kg/m<sup>2</sup>] = weight [kg] / (height [m])<sup>2</sup>
- Smoking status: Never smoker, Ex-smoker, Current smoker, Unknown
- Pack-Years
  - Pack-Years = packs a day \* years
- Indication of study drug: Chronic obstructive pulmonary disease (COPD), Other
- Chronic obstructive pulmonary disease (chronic bronchitis, emphysema) duration [years]

- If Month of first diagnosis of COPD is missing: COPD (chronic bronchitis, emphysema) duration = ([Years of first administration of Spiolto Respimat Years of first diagnosis of COPD])
- Severity: Mild, Moderate, Severe, Very severe
- Medical history: Yes, No, Unknown
  - Bronchial asthma: Yes, No, Unknown
  - Cardiac arrhythmia: Yes, No, Unknown
  - Ischaemic heart disease (coronary artery disease): Yes, No, Unknown
  - Cardiac failure (heart failure): Yes, No, Unknown
  - Cardiac arrest (resuscitation): Yes, No, Unknown
  - Cerebrovascular disorders, stroke: Yes, No, Unknown
  - Other cardiovascular disease: Yes, No, Unknown
  - Metabolic disorders: Yes, No, Unknown
  - Psychiatric disorders: Yes, No, Unknown
  - Renal and urinary disorders: Yes, No, Unknown
- Concomitant disease Yes, No, Unknown
  - Bronchial asthma: Yes, No, Unknown
  - Cardiac arrhythmia: Yes, No, Unknown
  - Ischaemic heart disease (coronary artery disease): Yes, No, Unknown
  - Cardiac failure (heart failure): Yes, No, Unknown
  - Cardiac arrest (resuscitation): Yes, No, Unknown
  - Cerebrovascular disorders, stroke: Yes, No, Unknown
  - Other cardiovascular disease: Yes, No, Unknown
  - Metabolic disorders: Yes, No, Unknown
  - Psychiatric disorders: Yes, No, Unknown
  - Renal and urinary disorders: Yes, No, Unknown
  - Renal function disorders: Yes, No, Unknown
  - Hepatic function disorders: Yes, No, Unknown
- COPD Assessment Test (CAT):
  - CAT score at baseline (each score and sum of 8 questions)
- Pulmonary Function Test (PFT): Baseline FEV<sub>1</sub> [L]
  - Baseline FEV<sub>1</sub> [L] post bronchodilator
  - Baseline FEV<sub>1</sub> [L] pre bronchodilator
  - Baseline %FEV<sub>1</sub> [%]
  - Baseline %FEV<sub>1</sub> [%] post bronchodilator
  - Baseline %FEV<sub>1</sub> [%] pre bronchodilator
  - Baseline FVC [L]
  - Baseline FVC [L] post bronchodilator
  - Baseline FVC [L] pre bronchodilator
  - Baseline %FVC [%]
  - Baseline %FVC [%] post bronchodilator
  - Baseline %FVC [%] pre bronchodilator
  - Baseline EFV<sub>1</sub>/FVC [%]
  - Baseline EFV<sub>1</sub>/FVC [%] post bronchodilator
  - Baseline EFV<sub>1</sub>/FVC [%] pre bronchodilator

TSAP for BI Trial No: 1237.34

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Note:

"post bronchodilator"; That fall under any of the following.

- Use of long-acting bronchodilator within 8 hours before PFT
- Use of long-acting bronchodilator (twice daily type) within 12 hours before PFT
- Use of long-acting bronchodilator (once daily type) within 24 hours before PFT "pre bronchodilator"; That fall under all of the following.
- Not use of long-acting bronchodilator within 8 hours before PFT
- Not use of long-acting bronchodilator (twice daily type) within 12 hours before PFT
- Not use of long-acting bronchodilator (once daily type) within 24 hours before PFT

note:% FEV<sub>1</sub> [%] = (FEV<sub>1</sub> [L]) / ( (0.036: if male, 0.022: if female)\*(height [cm]) - (0.028: if male, 0.022: if female)\*age - (1.178: if male, 0.005: if female) )\*100 %FVC [%] = (FVC [L]) / ( <math>(0.042: if male, 0.031: if female)\*(height [cm]) - (0.024: if male, 0.019: if female)\*age - (1.785: if male, 1.105: if female) )\*100 (Please refer (2).)

- Pregnancy: Yes, No, Unknown
- Previous medications: Yes, No, Unknown

Medication administered from 28 days before administration of Spiolto Respimat to 1 day before administration of Spiolto Respimat.

- Respiratory medication: Yes, No note: Respiratory medication = LAMA, LABA and/or ICS
- LAMA monotherapy: Yes, No
- LABA monotherapy: Yes, No
- ICS monotherapy: Yes, No
- ICS+LABA (free combination + fixed dose combination): Yes, No
- ICS+LAMA (free combination + fixed dose combination): Yes, No
- LAMA+LABA (free combination + fixed dose combination): Yes, No
- ICS+LAMA+LABA (free combination + fixed dose combination):Yes, No Other respiratory medication
- Theophylline: Yes, No
- Mucolytic: Yes, No
- Concomitant medications: Yes, No, Unknown
  - Respiratory medication: Yes, No

note: Respiratory medication = LAMA, LABA and/or ICS

- LAMA monotherapy: Yes, No
- LABA monotherapy: Yes, No
- ICS monotherapy: Yes, No
- ICS+LABA (free combination + fixed dose combination): Yes, No
- ICS+LAMA (free combination + fixed dose combination): Yes, No
- LAMA+LABA (free combination + fixed dose combination): Yes, No
- ICS+LAMA+LABA (free combination + fixed dose combination):Yes, No Other respiratory medication
- Theophylline: Yes, No
- Mucolytic: Yes, No
- Previous therapy: Yes, No, Unknown

• Concomitant therapy: Yes, No, Unknown

# Treatment exposure:

- Duration of Spiolto Respimat treatment [days] = (date of last treatment intake) (date of first intake) + 1
  - If after the data lock, Spiolto Respimat is ongoing and date of last treatment intake is missing: date of last treatment intake = Latest date in book
- Duration of Spiolto Respimat treatment class [weeks]: <= 4 weeks, 4 to <= 12 weeks, 12 to <=24 weeks, 24 to <=52 weeks, > 52 weeks.
  - Note: In terms of days <= 29days, 29 to <= 85days, 85 to <= 169, 169 to <= 365, >365

## 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENT(S)

For basic information on treatment in the study, please refer to NIS Protocol Section 4. The technical specification for treatment set-up is described in the Analysis Data Set (ADS) plan.

For safety analyses, data up to 21 days after last treatment intake during observation period will be considered as on treatment for AE.

#### 6.2 IMPORTANT PROTOCOL VIOLATIONS

The following table defines the different categories of important PVs. The final column describes which PVs will be used to exclude patients from the each patient analysis sets.

Observed PVs will be concluded as important or not important at report planning meetings before database lock at the latest.

Table 6.2:1 Important protocol violations

| Category / | | Description | Requirements | Method | Excluded from |
|---|---|---|---|---|---|
| Coo | de | | | | |
| A | | Entrance criteria not met | | | |
| | A1 | No COPD(chronic bronchitis, emphysema) | | Automated | Effectiveness |
| | A2 | Patient received Spiolto Respimat treatment before registration | See Previous Medication code: | Automated | Safety<br>Effectiveness |
| | A3 | Patients who have been enrolled this study before | | Manual | Safety<br>Effectiveness |
| | A4 | Patients who are participating in a clinical trial or registry. | | Manual | Safety<br>Effectiveness |
| В | | Contract | | | |
| | B1 | No valid site contract was available | | Manual | Safety<br>Effectiveness |
| C | | Trial medication | | | |
| | C1 | No treatment with Spiolto<br>Respimat | | Automated | Safety<br>Effectiveness |
| D | | Missing data | | | |
| | D1 | No patient visit after registration | See CRF "Administration status" | Automated | Safety<br>Effectiveness |
| | D2 | No CRF after registration | | Automated | Safety<br>Effectiveness |
| | D3 | No Effectiveness data | No Patient's Global Rating, no Physicians' global assessment and no available change value from baseline of CAT, FEV <sub>1</sub> and FVC. | Automated | Effectiveness |

#### 6.3 PATIENT SETS ANALYSED

The safety set and the effectiveness set are defined as follows. The safety set will be the basis of all demographic, baseline and safety analyses. Effectiveness analysis will be on basis of the effectiveness set.

- Safety set:
  - This patient set includes all patients who were documented to have taken at least one dose of Spiolto Respimat.
- Effectiveness set:

This patient set is a subset of the safety set that not received Spiolto Respimat patients before registration, and who have change value from baseline at least one CAT, FEV1 and FVC.

#### 6.5 POOLING OF CENTRES

This section is not applicable because centre/country is not included in the statistical model.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

If only year of date is non-missing, then missing date are imputed 01 JUL of reported year. Else if only year and month of date are non-missing, then missing date is imputed 15 of the reported month.

#### Safety:

Missing or incomplete AE dates are imputed according to BI standards (see "Handling of missing and incomplete AE dates"). (1)

#### Effectiveness:

Missing effectiveness data will not be imputed.

## 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

With regard to effectiveness and safety endpoints, the term "baseline" refers to the last observed measurement prior to administration of Spiolto Respimat. Observation on the same day as administration of Spiolto Respimat is "baseline".

Effectiveness analyses will be performed based on calculated visits as shown in Table 6.7: 1. If two or more data points of a patient fall into the same interval, the closest value to the planned day will be selected. If there are two observations which have the same difference in days to the planned day or if there are two observations on the same day, the first value will be used.

Table 6.7:1 Baseline, time windows and calculated visits

| | | Time window ( | Time window (actual days on treatment) |
|---|---|---|---|
| Week label | Planned days | Start | End |
| Baseline | 1 | The last observed measurement prior to or on administration of Spiolto Respimat | |
| Week4 | 29 | 2 | 57 |
| Week12 | 85 | 58 | 127 |
| Week24 | 169 | 128 | 267 |
| Week52 | 365 | 268 | End of study |

# 7. PLANNED ANALYSIS

For End-Of-Text (EoT) tables, the set of summary statistics is: N / Mean / SD / Min / Q1 / Median / Q3 / Max. For tables that are provided for endpoints with some extreme data, median, quartiles and percentiles should be preferred to mean, standard deviation, minimum and maximum.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group (unless otherwise specified, all patients in the respective patient set whether they have non-missing values or not). Percentages will be rounded to 2 decimal places. The category missing will be displayed only if there are actually missing values.

In addition, individual values on demographics, safety and effectiveness will be presented in subject data listings.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Concomitant diseases will be coded by the latest version of Medical Dictionary for Regulatory Activities (MedDRA). Frequency of patients will be summarized by system organ class (SOC) and preferred term (PT).

Concomitant medication will be coded by latest version of "Nihon-iyakuhinshu".

#### 7.3 TREATMENT COMPLIANCE

Compliance data is not collected in this study

# 7.4 PRIMARY ENDPOINT(S)

The analysis of the primary endpoint is described in Section 7.8.1.

#### 7.5 SECONDARY ENDPOINT(S)

The secondary endpoints will be used as stated in the NIS Protocol Section 9.7.3.

## 7.5.1 Key secondary endpoint(s)

TSAP for BI Trial No: 1237.34

This section is not applicable as no key secondary endpoint has been specified in the protocol.

# 7.5.2 (Other) Secondary endpoint(s)

This section is not applicable as no secondary endpoint has been specified in the protocol.

#### 7.7 EXTENT OF EXPOSURE

Only descriptive statistics are planned for this section of the report.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the treated set.

#### 7.8.1 Adverse events

Unless otherwise specified, the analyses of adverse events will be descriptive in nature. All analyses of AEs will be based on the number of patients with AEs and NOT on the number of AEs.

For further details on summarization of AE data, please refer to the guideline 'Analysis and Presentation of Adverse Event Data from Clinical Trials (1)

AE analyses will be carried out after integrating AE data from CRF and AE data from perceive system. In addition, AEs coded as "no adverse event" will not be included in the AE analyses.

The analysis of adverse events will be based on the concept of treatment emergent adverse events. That means that all adverse events occurring between first drug intakes till 21 days after last drug intake during observation period will be analysed. For details on the treatment definition, see Section 6.1.

An overall summary of adverse events will be presented.

The frequency of patients with AEs, ADRs, SAEs and SADRs will be summarised by primary system organ class and preferred term. Patients with 'priority survey items' according to the drug's Risk Management Plan will be summarised separately. The analysis of "priority survey items", "Important identified risks", "Important potential risks" will be conducted for AEs, ADRs.

It is created that table of patient with ADRs in each subgroup defined in Section 6.4. Not only the frequency but also the odds ratios are displayed.

In addition summaries for the time to onset of first episode for the ADRs will be tabulated, by duration (<= 4 week, 4 to <= 12 weeks, 12 to <=24 weeks, 24 to <=52 weeks, > 52), by primary system organ class and preferred term.

Adverse events leading to death and adverse events leading to discontinuation will be also summarised by treatment, primary system organ class and preferred term.

An ADR is defined as an AE for which either the investigator or the sponsor (or both) assess the causal relationship to Spiolto Respimat as "Yes". A SAE is defined as an AE for which either the investigator or the sponsor (or both) assess the seriousness either as "Serious".

The system organ classes will be sorted according to the standard sort order specified by EMA, preferred terms will be sorted by frequency (within system organ class).

The following AEs are detected on the basis of the Standardised MedDRA queries (SMQs) or Boehringer Ingelheim customised MedDRA query (BICMQ) (details are described in ADS plan).

Safety will be assessed by treatment exposure time adjusted incidence rate (n in 100 patient years) of ADRs.

#### Priority survey items

- Cardiovascular adverse events
- Anticholinergic-related adverse events
- Beta2 agonist-related events

#### Important identified risks

- Cardiac failure
- Atrial fibrillation and extra systoles
- Ileus, Angle closure glaucoma
- Anaphylaxis

#### Important potential risks

• Cardiac disorder (Myocardial ischaemia, Cardiac arrhythmia)

• Intubation and mortality related to asthma

## 7.8.2 Laboratory data

Only clinically relevant findings reported as AE will be analyzed as a part of AE analyses

# 7.8.3 Vital signs

Only clinically relevant findings reported as AE will be analysed as a part of AE analyses

# 7.8.4 ECG

Only clinically relevant findings reported as AE will be analyzed as a part of AE analyses

# **7.8.5** Others

No plan for other safety parameters.

Boehringer Ingelheim
TSAP for BI Trial No: 1237.34
Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8. **REFERENCES**

| 1 | 001-MCG-156: "Handling and summarization of adverse event data for clinical trial |
|---|---|
| | reports and integrated summaries", current version; IDEA for CON. |
| 2 | Annals of the Japanese Respiratory Society. 2001; 39: 1-17. |

TSAP for BI Trial No: 1237.34 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1237.34 
Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **10. HISTORY TABLE**

Table 10:1 History table

| Version | Date<br>(DD-MMM-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Final | 29 -Nov-2018 | | None | This is the final TSAP without any modification |